CLINICAL TRIAL: NCT05195749
Title: A Prospective, Phase II Study to Evaluate Safety of 101-PGC-005 ('005) for Moderate to Severe COVID-19 Disease Along With Standard of Care
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: 101 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGC-005-CP-101
Record Dates: First submitted 2022-01-11; First posted 2022-01-19 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: Glucocorticoids; Corticosteroids; Dexamethasone; Infectious disease; Cytokine storm
MeSH Terms: conditions — COVID-19; Communicable Diseases; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: 19 eligible patients will be enrolled to receive '005 + Standard of Care (SOC) and 10 patients will be enrolled to a control group receiving the SOC + placebo. The 1st open-label stage a 3+3+3 design will be implemented. 3 patients will receive 10mg '005 + SOC, 3 patients will receive 20mg '005 + SOC, and 3 patients will receive 30mg '005 + SOC. If no safety concerns are identified the 2nd stage will be initiated. All dose-escalation decisions will be based on previous cohort safety data, and doses will not be escalated unless 2 patients receiving the highest current dose have been observed for 24 hours post the 3rd dose. At the 2nd double blind stage neither the participants nor the investigator will know which treatment participants are receiving until the clinical trial is over. 20 patients will be enrolled and randomly allocated in a 1:1 ratio to the treatment (SOC + '005) or placebo group (SOC + placebo). The treatment dose will be chosen based on the 1st stage safety results.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, neither the participants nor the investigator is aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Patients (Experimental): Moderate to severe COVID-19 patients receiving SOC and '005.
  Interventions: Drug: 101-PGC-005 ('005) + SOC
- Control (Placebo Comparator): Moderate to severe COVID-19 patients receiving SOC and placebo.
  Interventions: Drug: Placebo + SOC

INTERVENTIONS:
Drug: 101-PGC-005 ('005) + SOC — Three consecutive days of '005 administration
  Arms: COVID-19 Patients
Drug: Placebo + SOC — Three consecutive days of placebo administration
  Arms: Control

SUMMARY:
In December 2019, a novel pneumonia caused by a previously unknown pathogen emerged in Wuhan, China. The pathogen was soon identified as a novel coronavirus (SARS-CoV-2), which is closely related to severe acute respiratory syndrome CoV (SARS-CoV) COVID-19, caused by the SARS-CoV-2 virus, leading to a major global public health threat. Many COVID-19 patients develop acute respiratory distress syndrome (ARDS) leading to death. The recent RECOVERY Trial demonstrated the success of dexamethasone in treating late-stage COVID-19 patients. However, use of dexamethasone increases mortality in the early stage of the disease, and dexamethasone is further limited because the therapeutic dose and duration is insufficient to safely and effectively treat most COVID-19 patients. As the majority of cells have glucocorticoid receptors to which dexamethasone binds, highly toxic doses would be needed to effectively treat COVID-19, which results in increased mortality as well as decreased natural immunity (via T-cell and other immune cell modulation). The investigational product 101-PGC-005 ('005) - a prodrug of dexamethasone that is targeted to only activated macrophages - will address the many safety and efficacy issues that limit dexamethasone. '005 can achieve much higher anti-inflammatory doses and avoid all undesirable immunosuppressive activities caused by standard dexamethasone administration, resulting in an even greater reduction in mortality among hospitalized patients and significantly reducing long term morbidity in patients who survive.

DETAILED DESCRIPTION:
This prospective Phase IIa study will evaluate the safety of '005 for moderate to severe COVID-19 disease along with Standard of Care (SOC) treatment. The Nineteen (19) eligible patients will be enrolled to receive '005 + SOC, 10 additional patients will be enrolled to a control group receiving the SOC together with placebo.

At the first open-label stage, 3+3+3 design will be implemented. Three (3) patients will be enrolled to receive 10mg '005 together with SOC, three (3) patients will receive 20mg'005 together with SOC, and three (3) patients will receive 30mg '005 together with SOC if no safety concerns are identified the second stage will be initiated.

At the second double blind stage neither the participants nor the investigator will know which treatment participants are receiving until the clinical trial is over [20 patients will be enrolled and randomly allocated in a 1:1 ratio to the treatment (SOC +'005) or placebo group (SOC + placebo)]. The treatment dose will be chosen based on the first stage safety results.

NOTE: '005 will be administered daily for three (3) consecutive days starting from the day of enrollment.

Standard of Care will be administered as long as required, per Investigator's judgment, institutional practice, or local, national, or international guidelines for COVID-19 management.

A screening period of up to 7 days (Day-7 to Day-1) prior to enrollment will be followed by a study period of 28 days. Patients will be administered '005 daily from Day-1 to Day 3.

Total duration of study participation will not exceed 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to provide voluntary written informed consent and to follow the protocol specific requirements.
* Male or female patients over 18 years old.
* Patients with positive RT-PCR test for SARS-CoV-2 in nasopharyngeal or oropharyngeal swabs (sample collected within 7 days prior to enrollment) who are admitted or being admitted to the hospital for a primary diagnosis of COVID-19.
* In the case of female patients of child-bearing potential, a negative blood pregnancy test prior to beginning the therapy.
* Patients intended to be hospitalized to receive SOC including dexamethasone treatment for COVID-19.

Exclusion Criteria:

Exclusion Criteria:

* Patients with evidence of other serious infections.
* Malignancy.
* Background disease which, in the opinion of the investigator prevents the patient from participating in the study such as:

  * Presence of serious chronic infectious.
  * A condition resulting in immunodeficiency.
  * Participants with glucose levels upon admission ≥ 250 mg/dL
  * Acute psychosis
* Patients in a critical stage of COVID-19 disease that require mechanical ventilation.
* Pregnant and lactating women.
* Patients that are currently or have participated in other clinical studies with investigational drug, biological agent, or device within 1 month or within 5 half-lives (of the drug/biologic) prior to enrollment (whichever is longer).
* Patient currently receiving chemotherapy or immunosuppressive agents not including dexamethasone within 30 days before the screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 2. | At day 2
  Evaluate the incidence of steroid-induced hyperglycemia Fasting Plasma Glucose (FPG).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 3. | At day 3
  Evaluate the incidence of steroid-induced hyperglycemia Fasting Plasma Glucose (FPG).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 4. | At day 4
  Evaluate the incidence of steroid-induced hyperglycemia Fasting Plasma Glucose (FPG).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 10. | At day 10
  Evaluate the incidence of steroid-induced hyperglycemia Fasting Plasma Glucose (FPG).

SECONDARY OUTCOMES:
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 2. | At day 2
  Evaluate the incidence of vital signs abnormality (i.e., pulse, oxygen saturation and blood pressure).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 3. | At day 3
  Evaluate the incidence of vital signs abnormality (i.e., pulse, oxygen saturation and blood pressure).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 4. | At day 4
  Evaluate the incidence of vital signs abnormality (i.e., pulse, oxygen saturation and blood pressure).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment at day 10. | At day 10
  Evaluate the incidence of vital signs abnormality (i.e., pulse, oxygen saturation and blood pressure).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 28
  Evaluate the incidence of vital signs abnormality (i.e., pulse, oxygen saturation and blood pressure).
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 2
  Evaluate the incidence of clinically significant changes in the blood CBC, and biochemistry.
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 3
  Evaluate the incidence of clinically significant changes in the blood CBC, and biochemistry.
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 4
  Evaluate the incidence of clinically significant changes in the blood CBC, and biochemistry.
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 10
  Evaluate the incidence of clinically significant changes in the blood CBC, and biochemistry.
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At day 28
  Evaluate the incidence of clinically significant changes in the blood CBC, and biochemistry.
To assess the safety of '005 in moderate to severe COVID-19 patients with Standard of Care treatment. | At 28 days
  Evaluate incidence of Adverse Events/Serious Adverse Events (AEs/SAEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) thru the study.
The 28 days discharge rate. | At 28 days
  Comparison of 28 days discharge rate.
COVID-19 severity improvement by MOH COVID-19 severity scale while in hospital, and at days 10 and 28 if discharged. | At 10 days
  COVID-19 severity improvement by MOH COVID-19 severity scale while in hospital, and at days 10 and 28 if discharged .
COVID-19 severity improvement by MOH COVID-19 severity scale while in hospital, and at days 10 and 28 if discharged. | At 28 days
  COVID-19 severity improvement by MOH COVID-19 severity scale while in hospital, and at days 10 and 28 if discharged .
Reduction in inflammatory blood markers. | At 10 days
  Reduction in CRP, or Ferritin levels at days 10 and 28.
Reduction in inflammatory blood markers. | At 28 days
  Reduction in CRP, or Ferritin levels at days 10 and 28.
Improvement of COVID-19 symptoms. | At day 28
  Improvement in 1 or more COVID-19 symptoms severity from baseline (temperature, rate PaO2/FiO2, Mechanical ventilation or not mechanical ventilation) at days 10 or 28.
Improvement of COVID-19 symptoms. | At day 10
  Improvement in 1 or more COVID-19 symptoms severity from baseline (temperature, rate PaO2/FiO2, Mechanical ventilation or not mechanical ventilation) at days 10 or 28.
Time to Saturation ≥94% on Room Air | At day 10
  Time to Saturation ≥94% on Room Air at day 10
Time to Saturation ≥94% on Room Air | At day 28
  Time to Saturation ≥94% on Room Air at day 28.
Blood evaluation for '005 PK. | At day 1: at baseline 30 min, 1, 2, 4, 5, 6, 8 and 24hr post dose
  Evaluation of '005 kinetics in the blood at Day 1: at baseline 30 min, 1, 2, 4, 5, 6, 8 and 24hr post dose
Blood evaluation for '005 PK. | At day 3: at baseline 30 min, 1, 2, 4, 5, 6, 8 and 24hr post dose
  Evaluation of '005 kinetics in the blood at Day 3: at baseline 30 min, 1, 2, 4, 5, 6, 8 and 24hr post dose
Changes from baseline in pro-inflammatory cytokines and Lymphocyte subtypes. | At day 4
  Changes from baseline in pro-inflammatory cytokines and Lymphocyte subtypes at Day 4 and 10.
Changes from baseline in pro-inflammatory cytokines and Lymphocyte subtypes. | At day 10
  Changes from baseline in pro-inflammatory cytokines and Lymphocyte subtypes at Day 4 and 10.
Correlation with pro-inflammatory cytokines and change in COVID-19 symptoms | At day 4
  Correlation with pro-inflammatory cytokines and change in COVID-19 symptoms at Day 4.
Correlation with pro-inflammatory cytokines and change in COVID-19 symptoms | At day 10
  Correlation with pro-inflammatory cytokines and change in COVID-19 symptoms at Day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Khetam Hussein, MD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- The COVID-19 Unit, Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No